CLINICAL TRIAL: NCT04673175
Title: A Pilot Study of Ceftolozane-Tazobactam in Conjunction With Rapid Molecular Diagnosis for Directed Treatment of Pseudomonas Aeruginosa Bacteremia and Pneumonia in Patients With Hematological Malignancies and Hematopoietic Stem Cell Transplantation
Brief Title: Ceftolozane-Tazobactam for Directed Treatment of Pseudomonas Aeruginosa Bacteremia and Pneumonia in Patients With Hematological Malignancies and Hematopoietic Stem Cell Transplantation
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to slow accrual.
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-11021048
Record Dates: First submitted 2020-12-04; First posted 2020-12-17 (Actual); Results first posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Pneumonia; Hematologic Malignancy; Pseudomonas Aeruginosa Infection; Bacteremia; Hematopoietic Stem Cell Transplant (HSCT)
Keywords: Pseudomonas Aeruginosa; Pneumonia; Hematologic Malignancy; Ceftolozane-Tazobactam; Zerbaxa; Stem Cell Transplant Recipients; Immunocompromised Hosts; Gram-Negative Bacterial Infections
MeSH Terms: conditions — Pneumonia; Hematologic Neoplasms; Pseudomonas Infections; Bacteremia; Gram-Negative Bacterial Infections | interventions — ceftolozane, tazobactam drug combination

STUDY DESIGN:
Intervention Model Description: The study includes two groups analyzed in parallel: (1) a prospective treatment arm in which participants receive ceftolozane-tazobactam for Pseudomonas aeruginosa infection, and (2) a historical control arm consisting of patients previously treated with standard-of-care anti-pseudomonal therapy. Historical controls are identified retrospectively and are not prospectively assigned or treated under this protocol.
Masking Description: This is an open-label study. No parties are masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ceftolozane-Tazobactam (Prospective Treatment Arm) (Experimental): Participants prospectively enrolled in the study received ceftolozane-tazobactam intravenously every 8 hours for approximately 10 to 14 days, with treatment extended up to 21 days if infection persisted or recurred. Outcomes for this arm were assessed according to the protocol's primary and secondary endpoints.
  Interventions: Drug: Ceftolozane / Tazobactam Injection
- Historical Control (Standard of Care Prior to Study) (No Intervention): This arm consists of historical control patients with documented Pseudomonas aeruginosa bacteremia and/or pneumonia who received standard-of-care antimicrobial therapy prior to initiation of this study. These patients were included retrospectively for comparative analyses of selected primary and secondary endpoints. No study interventions were administered to this arm.

INTERVENTIONS:
Drug: Ceftolozane / Tazobactam Injection — Zerbaxa (ceftolozane/tazobactam) for injection is supplied as a white to yellow sterile powder for reconstitution in single-use vials; each vial contains 1 g ceftolozane (equivalent to 1.147 g of ceftolozane sulfate) and 0.5 g tazobactam (equivalent to 0.537 g of tazobactam sodium).
  Arms: Ceftolozane-Tazobactam (Prospective Treatment Arm)

SUMMARY:
The goal of this clinical trial is to learn whether the antibiotic ceftolozane-tazobactam works to treat serious Pseudomonas aeruginosa infections in people with blood cancers or who received a stem cell transplant. The main question it aims to answer is whether participants reach clinical success 30 days after the infection is first found. Clinical success means the person is alive, their infection symptoms are improving, and the infection has not returned.

Participants will receive ceftolozane-tazobactam through a vein every 8 hours for 10 to 14 days. Treatment may continue for up to 21 days if the infection is not improving or keeps coming back. The infection is diagnosed using the hospital's standard rapid molecular tests, which help confirm Pseudomonas aeruginosa quickly so treatment can begin right away.

Researchers will follow participants during their hospital stay and check on them around 30 and 60 days to see how well the treatment worked. The study will also look at how long it takes for the infection to clear, how long participants stay in the hospital or intensive care unit, and whether the bacteria become resistant to antibiotics.

In addition to the prospective ceftolozane-tazobactam group, the study includes a historical control group made up of patients with similar infections who were treated in the past with standard anti-pseudomonal antibiotics (such as cefepime, ceftazidime, piperacillin-tazobactam, or meropenem). Data from these historical controls are collected by chart review and analyzed alongside the prospective group to compare outcomes. Historical controls do not receive study-directed treatment and are not actively enrolled under this protocol.

ELIGIBILITY:
Eligibility Criteria

Inclusion Criteria

* Presence of a hematologic malignancy or a history of hematopoietic stem cell transplantation
* Identification of Pseudomonas aeruginosa by rapid molecular diagnostic testing from a positive blood culture or from a respiratory sample in the setting of radiologically documented pneumonia with compatible clinical symptoms
* Age 18 years or older
* Ability of the participant or legally authorized representative to provide informed consent

Exclusion Criteria

* Receipt of more than 72 hours of non-study anti pseudomonal therapy for the infection being treated
* Known anaphylactic hypersensitivity or allergic reaction to cephalosporins
* History of a Pseudomonas aeruginosa isolate with a ceftolozane or tazobactam MIC greater than 4 micrograms per milliliter
* Polymicrobial aerobic Gram negative infection, as determined by the infectious diseases research team
* Hemodialysis, continuous renal replacement therapy, or creatinine clearance less than 15 milliliters per minute
* Expected mortality within 48 hours of screening

Eligibility Criteria for Historical Controls

Inclusion Criteria

* Presence of a hematologic malignancy or a history of hematopoietic stem cell transplantation
* Identification of Pseudomonas aeruginosa associated with bacteremia and or pneumonia
* Age 18 years or older
* Survival greater than 48 hours after initiation of anti pseudomonal therapy for Pseudomonas aeruginosa bacteremia and or pneumonia

Exclusion Criteria

* Known anaphylactic hypersensitivity or allergic reaction to cephalosporins
* History of a Pseudomonas aeruginosa isolate with a ceftolozane or tazobactam MIC greater than 4 micrograms per milliliter
* Polymicrobial aerobic Gram negative infection, as determined by the infectious diseases research team
* Hemodialysis, continuous renal replacement therapy, or creatinine clearance less than 15 milliliters per minute

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2025-03-16 (Actual); Study Completion 2025-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Markus Plate, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Satlin MJ, Walsh TJ. Multidrug-resistant Enterobacteriaceae, Pseudomonas aeruginosa, and vancomycin-resistant Enterococcus: Three major threats to hematopoietic stem cell transplant recipients. Transpl Infect Dis. 2017 Dec;19(6):10.1111/tid.12762. doi: 10.1111/tid.12762. Epub 2017 Oct 25. PMID 28815897
- [Background] Freifeld AG, Bow EJ, Sepkowitz KA, Boeckh MJ, Ito JI, Mullen CA, Raad II, Rolston KV, Young JA, Wingard JR; Infectious Diseases Society of America. Clinical practice guideline for the use of antimicrobial agents in neutropenic patients with cancer: 2010 update by the infectious diseases society of america. Clin Infect Dis. 2011 Feb 15;52(4):e56-93. doi: 10.1093/cid/cir073. PMID 21258094
- [Background] Nguyen L, Garcia J, Gruenberg K, MacDougall C. Multidrug-Resistant Pseudomonas Infections: Hard to Treat, But Hope on the Horizon? Curr Infect Dis Rep. 2018 Jun 6;20(8):23. doi: 10.1007/s11908-018-0629-6. PMID 29876674
- [Background] Kaye KS, Pogue JM. Infections Caused by Resistant Gram-Negative Bacteria: Epidemiology and Management. Pharmacotherapy. 2015 Oct;35(10):949-62. doi: 10.1002/phar.1636. PMID 26497481
- [Background] Munita JM, Aitken SL, Miller WR, Perez F, Rosa R, Shimose LA, Lichtenberger PN, Abbo LM, Jain R, Nigo M, Wanger A, Araos R, Tran TT, Adachi J, Rakita R, Shelburne S, Bonomo RA, Arias CA. Multicenter Evaluation of Ceftolozane/Tazobactam for Serious Infections Caused by Carbapenem-Resistant Pseudomonas aeruginosa. Clin Infect Dis. 2017 Jul 1;65(1):158-161. doi: 10.1093/cid/cix014. PMID 28329350
- [Background] Gallagher JC, Satlin MJ, Elabor A, Saraiya N, McCreary EK, Molnar E, El-Beyrouty C, Jones BM, Dixit D, Heil EL, Claeys KC, Hiles J, Vyas NM, Bland CM, Suh J, Biason K, McCoy D, King MA, Richards L, Harrington N, Guo Y, Chaudhry S, Lu X, Yu D. Ceftolozane-Tazobactam for the Treatment of Multidrug-Resistant Pseudomonas aeruginosa Infections: A Multicenter Study. Open Forum Infect Dis. 2018 Oct 31;5(11):ofy280. doi: 10.1093/ofid/ofy280. eCollection 2018 Nov. PMID 30488041
- [Background] Petraitis V, Petraitiene R, Naing E, Aung T, Thi WP, Kavaliauskas P, Win Maung BB, Michel AO, Ricart Arbona RJ, DeRyke AC, Culshaw DL, Nicolau DP, Satlin MJ, Walsh TJ. Ceftolozane-Tazobactam in the Treatment of Experimental Pseudomonas aeruginosa Pneumonia in Persistently Neutropenic Rabbits: Impact on Strains with Genetically Defined Mechanisms of Resistance. Antimicrob Agents Chemother. 2019 Aug 23;63(9):e00344-19. doi: 10.1128/AAC.00344-19. Print 2019 Sep. PMID 31235620

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Prospective participants for the ceftolozane-tazobactam arm were recruited at a single academic tertiary care hospital among adults with hematologic malignancies or hematopoietic stem cell transplant and documented Pseudomonas aeruginosa bacteremia or pneumonia between January 2023 and February 2025. Historical controls were identified retrospectively from the same institution.
Pre-assignment Details: A total of 17 consent events occurred among 16 unique participants. Per protocol, one participant was eligible for re-enrollment after developing a separate Pseudomonas aeruginosa infection and received study treatment during both enrollments. For statistical analyses, this participant was counted once to avoid bias. Analyses therefore summarize outcomes for 16 unique treated participants.
Period: Overall Study
Arm/Group | Ceftolozane-Tazobactam (Prospective Treatment Arm) | Historical Control (Standard of Care Prior to Study)
Started | 16 (One participant was intentionally re-enrolled per protocol for a second, distinct Pseudomonas aeruginosa infection. Although this individual consented and received study treatment twice, they are counted once in Participant Flow to reflect the number of unique participants assigned to the prospective treatment arm.) | 48
Completed (All 16 unique prospective participants and all 48 historical controls were included in the final analysis datasets. The duplicate prospective enrollment was counted once.) | 16 | 48
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were summarized for 16 unique prospective participants and 48 historical controls, matching the numbers in Participant Flow. The participant who was re-enrolled for a second Pseudomonas aeruginosa infection is counted once in the baseline tables, consistent with the analysis datasets.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ceftolozane-Tazobactam (Prospective Treatment Arm) | Historical Control (Standard of Care Prior to Study) | Total
Number analyzed (Participants) | 16 | 48 | 64
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 68.5 [64 to 71.5] | 66 [56 to 74.5] | 67 [58.5 to 73.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 23 | 24
  Male | 15 | 25 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 5 | 5
  Not Hispanic or Latino | 15 | 35 | 50
  Unknown or Not Reported | 1 | 8 | 9
Infection Type at Index Pseudomonas Infection [Count of Participants; unit: Participants] — Infection type at baseline at the time of the index Pseudomonas aeruginosa culture. Participants with both bacteremia and pneumonia were categorized under bacteremia. This variable was used for matching between the prospective arm and historical controls.
  Participants
    Bacteremia | 13 | 39 | 52
    Pneumonia | 3 | 9 | 12
Neutropenia Status at Index Pseudomonas Infection [Count of Participants; unit: Participants] — Neutropenia status at baseline was defined as an absolute neutrophil count (ANC) or white blood cell count below 0.5 × 10⁹/L at the time of the index Pseudomonas aeruginosa culture. This variable was used for matching between the prospective cohort and historical controls.
  Participants
    Neutropenic | 7 | 21 | 28
    Not Neutropenic | 9 | 27 | 36
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 0 | 0
  Race: Asian | 1 | 3 | 4
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Race: Black or African American | 1 | 7 | 8
  Race: White | 14 | 27 | 41
  Race: Other combinations not described | 0 | 9 | 9
  Race: Decline to answer | 0 | 2 | 2
Hematologic Malignancy Type [Number; unit: Participants] — Hematologic malignancy diagnoses present at the time of the index infection. Some participants had more than one underlying hematologic malignancy; therefore, individual participants may be counted in more than one category. Counts reflect diagnosis prevalence and are not mutually exclusive.
  Participants
    Acute myeloid leukemia | 8 | 18 | 26
    Acute lymphoblastic leukemia | 1 | 4 | 5
    Chronic leukemia | 3 | 3 | 6
    Non-Hodgkin's lymphoma | 3 | 14 | 17
    Multiple myeloma | 1 | 7 | 8
    Myelodysplastic Syndromes | 4 | 5 | 9
Hematopoietic cell transplant recipient [Count of Participants; unit: Participants] — Indicates whether participants had undergone any hematopoietic cell transplant (autologous, allogeneic, or both) before the index Pseudomonas aeruginosa infection. "Yes" includes participants with prior autologous, allogeneic, or both transplant types.
  Participants
    Yes | 10 | 18 | 28
    No | 6 | 30 | 36
Pitt Bacteremia Score [Median (Inter-Quartile Range); unit: score on a scale] — A validated severity-of-illness score ranging from 0 to 14, with higher scores indicating greater acute illness severity. Scores were assessed at the time of index culture collection and are reported as median and interquartile range.
  score on a scale | 0.5 [0 to 1] | 1 [0 to 2] | 1 [0 to 2]
Age-adjusted Charlson Comorbidity Index [Median (Inter-Quartile Range); unit: score on a scale] — A validated comorbidity score ranging from 0 to 37, with higher scores indicating greater comorbidity burden and mortality risk. Scores were assessed at the time of index culture collection and are reported as median and interquartile range.
  score on a scale | 6 [4 to 7] | 5 [4 to 7] | 5 [4 to 7]

OUTCOME MEASURES:

1. Primary Outcome: Clinical Success at Day 30
Description: Clinical success 30 days after collection of the index culture. Clinical success is defined as meeting all of the following criteria at that time point: survival; resolution or near resolution of baseline clinical manifestations, including fever, hypoxia, and signs or symptoms of sepsis; and absence of recurrent infection due to Pseudomonas aeruginosa or persistent infection despite more than 7 days of anti-pseudomonal therapy.
Time Frame: 30 days after collection of the index culture
Population: Outcome measures were summarized for 16 unique prospective participants and 48 historical controls, matching the numbers in Participant Flow. The participant who was re-enrolled for a second Pseudomonas aeruginosa infection is counted once for this measure, consistent with the analysis datasets.
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftolozane-Tazobactam (Prospective Treatment Arm) | Historical Control (Standard of Care Prior to Study)
Number analyzed (Participants) | 16 | 48
Participants
  Clinical Success | 12 | 30
  Clinical Failure | 4 | 18
Statistical Analysis 1: Comparison: Ceftolozane-Tazobactam (Prospective Treatment Arm) vs Historical Control (Standard of Care Prior to Study); Comparison of the proportion of participants with clinical success at Day 30 between the prospective ceftolozane-tazobactam arm and matched historical controls; Test type: Superiority; p = 0.40, Chi-squared; Two-sided Pearson chi-squared test comparing the prevalence of clinical success between arms

2. Secondary Outcome: Survival at Day 30
Description: Survival status 30 days after initiation of anti-pseudomonal therapy for the index infection, assessed by chart review or phone contact.
Time Frame: 30 days after initiation of anti-pseudomonal therapy for the index infection
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftolozane-Tazobactam (Prospective Treatment Arm) | Historical Control (Standard of Care Prior to Study)
Number analyzed (Participants) | 16 | 48
Participants
  Alive | 15 | 35
  Deceased | 1 | 13

3. Secondary Outcome: Survival at Day 60
Description: Survival status 60 days after initiation of anti-pseudomonal therapy for the index infection, assessed by chart review or phone contact.
Time Frame: 60 days after initiation of anti-pseudomonal therapy for the index infection
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftolozane-Tazobactam (Prospective Treatment Arm) | Historical Control (Standard of Care Prior to Study)
Number analyzed (Participants) | 16 | 48
Participants
  Alive | 13 | 28
  Deceased | 3 | 20

4. Secondary Outcome: Time to Resolution of Bacteremia
Description: Time (days) from the index positive blood culture for Pseudomonas aeruginosa to bacteremia resolution. Resolution was defined as the date of the first of two consecutive negative blood cultures obtained after the index culture. Participants without follow-up blood cultures were excluded from this analysis.
Time Frame: From index culture collection up to 60 days
Population: Analysis limited to participants with Pseudomonas aeruginosa bacteremia who had follow-up blood cultures after the index culture. Participants without follow-up blood cultures were excluded from this outcome. One participant in the prospective cohort was re-enrolled for a second Pseudomonas aeruginosa infection and is counted once for this measure, consistent with the analysis datasets.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Ceftolozane-Tazobactam (Prospective Treatment Arm) | Historical Control (Standard of Care Prior to Study)
Number analyzed (Participants) | 13 | 38
Days | 2 [1 to 2] | 1 [1 to 2]

5. Secondary Outcome: Length of Hospital Stay
Description: Total number of days hospitalized for the admission during which the index Pseudomonas aeruginosa infection is treated, measured beginning on the date of index culture collection and obtained from the Hospitalization Status Assessment.
Time Frame: From index culture collection through discharge from the hospital admission for the index infection (up to 60 days)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Ceftolozane-Tazobactam (Prospective Treatment Arm) | Historical Control (Standard of Care Prior to Study)
Number analyzed (Participants) | 16 | 48
Days | 17.5 [12 to 38] | 17 [12.5 to 25.5]

6. Secondary Outcome: Emergence of Ceftolozane-tazobactam Resistant Isolates
Description: Occurrence of Pseudomonas aeruginosa isolates that newly demonstrate resistance to ceftolozane-tazobactam on antimicrobial susceptibility testing after initiation of therapy for the index infection.
Time Frame: From index culture collection up to 60 days
Population: Assessed only among participants who received ceftolozane-tazobactam. Historical controls were not analyzed (0 participants) because they did not receive ceftolozane-tazobactam. One participant in the prospective cohort was re-enrolled for a second Pseudomonas aeruginosa infection and is counted once for this measure, consistent with the analysis datasets.
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftolozane-Tazobactam (Prospective Treatment Arm) | Historical Control (Standard of Care Prior to Study)
Number analyzed (Participants) | 16 | 0
Participants
  Emergence of ceftolozane-tazobactam resistant isolate | 0 |
  No emergence of ceftolozane-tazobactam resistant isolate | 16 |

7. Secondary Outcome: Time to Appropriate Therapy
Description: Time (in hours) from index culture collection for the index Pseudomonas aeruginosa infection to initiation of an anti-pseudomonal agent deemed appropriate based on antimicrobial susceptibility results.
Time Frame: From index culture collection up to 60 days
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Ceftolozane-Tazobactam (Prospective Treatment Arm) | Historical Control (Standard of Care Prior to Study)
Number analyzed (Participants) | 16 | 48
Hours | 1 [0 to 5.5] | 3 [0 to 22]

8. Secondary Outcome: Resolution of Baseline Clinical Manifestations
Description: Resolution or near resolution of baseline fever, hypoxia, or signs and symptoms of sepsis related to the index infection at 30 days after index culture collection, as assessed by physical examination findings and clinical documentation.
Time Frame: 30 days after collection of the index culture
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftolozane-Tazobactam (Prospective Treatment Arm) | Historical Control (Standard of Care Prior to Study)
Number analyzed (Participants) | 16 | 48
Participants
  Resolution or near resolution achieved | 14 | 33
  Resolution or near resolution not achieved | 2 | 15

9. Secondary Outcome: Modifications to Initial Antimicrobial Therapy
Description: Number of participants with any modification to the initial study-directed anti-pseudomonal regimen for the index infection, defined as either (1) discontinuation of ceftolozane-tazobactam with switch to another anti-pseudomonal agent or (2) addition of another anti-pseudomonal antibiotic during the treatment course. Outpatient levofloxacin was not considered a modification.
Time Frame: From initiation of study ceftolozane-tazobactam therapy through end of study-directed anti-pseudomonal treatment (up to 21 days)
Population: Assessed only among participants who received study-directed ceftolozane-tazobactam. Historical controls were not analyzed (0 participants) because they did not receive ceftolozane-tazobactam. One participant in the prospective cohort was re-enrolled for a second Pseudomonas aeruginosa infection and is counted once for this measure, consistent with the analysis datasets.
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftolozane-Tazobactam (Prospective Treatment Arm) | Historical Control (Standard of Care Prior to Study)
Number analyzed (Participants) | 16 | 0
Participants
  Modification to initial regimen | 3 |
  No modification to initial regimen | 13 |

10. Secondary Outcome: Emergence of Other Bacteria During Therapy
Description: Identification of new bacterial pathogens identified in blood cultures during study-directed ceftolozane-tazobactam treatment for the index infection.
Time Frame: From initiation of study ceftolozane-tazobactam therapy through end of ceftolozane-tazobactam treatment (up to 21 days)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftolozane-Tazobactam (Prospective Treatment Arm) | Historical Control (Standard of Care Prior to Study)
Number analyzed (Participants) | 16 | 0
Participants
  New bacterial pathogen identified | 0 |
  No new bacterial pathogen identified | 16 |

11. Secondary Outcome: Number of Days on Ventilator
Description: Total number of days requiring invasive mechanical ventilation during the index admission, measured beginning on the date of index culture collection and abstracted from the medical record.
Time Frame: From index culture collection through discharge from the hospital admission for the index infection (up to 60 days)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Ceftolozane-Tazobactam (Prospective Treatment Arm) | Historical Control (Standard of Care Prior to Study)
Number analyzed (Participants) | 16 | 48
Days | 0 [0 to 0] | 0 [0 to 0]

12. Secondary Outcome: ICU Length of Stay
Description: Total number of days spent in an intensive care unit during the index admission, measured beginning on the date of index culture collection and obtained from the Hospitalization Status Assessment.
Time Frame: From index culture collection through discharge from the hospital admission for the index infection (up to 60 days)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Ceftolozane-Tazobactam (Prospective Treatment Arm) | Historical Control (Standard of Care Prior to Study)
Number analyzed (Participants) | 16 | 48
Days | 0 [0 to 1] | 0 [0 to 2.5]

ADVERSE EVENTS:
Time Frame: From index culture collection through 60 days after initiation of anti-pseudomonal therapy (up to 60 days)
Description: SAEs were collected prospectively for participants receiving ceftolozane-tazobactam and classified per CTCAE v5.0. Only SAEs and deaths were systematically assessed; non-serious AEs were not collected. The participant who was re-enrolled for a second Pseudomonas aeruginosa infection episode is counted once for adverse event reporting purposes, consistent with the analysis datasets. AEs and SAEs for historical controls were not systematically collected, except for all-cause mortality.
Arm/Group | Ceftolozane-Tazobactam (Prospective Treatment Arm) | Historical Control (Standard of Care Prior to Study)
All-Cause Mortality (participants affected / at risk) | 3/16 | 20/48
Serious Adverse Events (participants affected / at risk) | 5/16 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ceftolozane-Tazobactam (Prospective Treatment Arm) (N=16) | Historical Control (Standard of Care Prior to Study) (N=0)
Suspected Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA — Grade 3 suspected aspiration following central venous catheter placement, associated with dysphagia after intubation. Required ICU transfer and escalation of respiratory support. Not related to study drug.
Graft-versus-host disease exacerbation (Immune system disorders) | 1 (1) | NA — Grade 3 worsening graft-versus-host disease attributed to donor lymphocyte infusion. Managed with immunosuppressive therapy escalation. Not related to study drug.
Pseudomonas aeruginosa bacteremia (Infections and infestations) | 1 (1) | NA — Grade 3 bacteremia associated with progression of bacterial pneumonia and respiratory decompensation, requiring ICU transfer. Not related to study drug.
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA — Grade 5 acute respiratory failure secondary to bacterial pneumonia and respiratory decompensation. Event resulted in death. Not related to study drug.
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | NA — Grade 3 febrile neutropenia following recent chemotherapy, requiring hospitalization. Not related to study drug.
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA — Grade 5 respiratory failure in the setting of progressive lymphoma and multiple infections, resulting in death. Not related to study drug.
Cytomegalovirus viremia (Infections and infestations) | 1 (1) | NA — Grade 4 CMV viremia requiring intravenous antiviral therapy. Viral load improved with treatment. Not related to study drug.
Death (General disorders) | 1 (1) | NA — Death occurred while hospitalized at an outside facility for complications of acute myeloid leukemia. The patient was transitioning to home hospice. Limited external medical records were available. Not related to study drug.

LIMITATIONS AND CAVEATS:
Limitations of this study include the lack of randomization between patients that received ceftolozane-tazobactam and alternative therapies, which creates the potential for confounding. Also, the modest sample size limited the statistical power to detect difference between groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-09): https://cdn.clinicaltrials.gov/large-docs/75/NCT04673175/Prot_SAP_000.pdf